CLINICAL TRIAL: NCT00323024
Title: An Open-Label, Dose-Determination Safety, Tolerability, and Activity Study of Inhaled NX1011 in Patients With Pulmonary Arterial Hypertension
Brief Title: Dose Determination Safety and Activity Study of Inhaled NX1011 to Treat Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NITROX, LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX1011:201
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2006-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Pulmonary Hypertension; Idiopathic PAH; PH associated with connective tissue disease (CTD); PH associated with interstitial lung disease (ILD); PH associated with congestive heart failure (CHF); PH associated with chronic obstructive pulmonary disease (COPD)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

INTERVENTIONS:
Drug: NX1011

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose of inhaled NX1011 for the treatment of pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Patient must either:

  * meet the PAH diagnostic criteria at Screening (based on a documented history of diagnosis as outlined in the American College of Chest Physicians [ACCP] 2004 Evidence-Based Clinical Practices Guidelines)15; or
  * have elevated pulmonary pressure with a suspected PAH diagnosis based on a clinical referral at Screening for a RHC.
* Patient must have PAH as defined by a mean pulmonary artery pressure (PAP) > 25 mmHg.
* Patient must have symptoms of pulmonary hypertension (PH) according to the World Health Organization (WHO) Functional Classification of Pulmonary Hypertension Class II through IV.
* Patient must consent to, be able to tolerate, and have adequate venous and arterial access for Swan-Ganz catheterization (SGC) and an arterial line.

Exclusion Criteria:

* Clinically significant right-to-left intracardiac shunts based on Doppler echocardiography with bubble study.
* History of pulmonary veno-occlusive disease or clinically significant aortic or mitral stenosis.
* History of sustained ventricular tachycardia (VT-S) or ventricular fibrillation (VF) and cardiac arrest, or presence of atrial fibrillation.
* Active cardiac disease meeting the following criteria:

  * Patient with elevated pulmonary capillary wedge pressures (PCWPs) > 25 mmHg.
  * Patient with a history of myocardial infarction or coronary intervention within the last 60 days.
  * Patient with a history of pacemaker, cardiac defibrillator, or biventricular pacemaker insertion within 4 weeks of Baseline.
  * Patient who cannot be withdrawn from nitrate therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2006-09; Study Completion 2007-05

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and activity of inhalation therapy with NX1011 based on right heart catheterization (RHC) measures, pulse oximetry, and hemodynamic response
To establish maximum tolerated dose (MTD) levels of NX1011 based on predefined criteria for dose-limiting toxicity (DLT)
To qualify the delivery apparatus
To generate descriptive data on the concentration-response relationship in order to choose a range of concentrations (e.g., low, medium, high) for the follow-up, fixed-dose, placebo-controlled study
To summarize correlation data between echocardiography and RHC measures with respect to activity and methemoglobin levels documented via the visible light spectroscopy

SECONDARY OUTCOMES:
To summarize correlation data between echocardiography and RHC measures with respect to activity and methemoglobin levels documented via the visible light spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Victoria A Christian, Study Director — NITROX, LLC
Locations (6):
- United States (6):
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of California, San Diego Medical Center, La Jolla, California
  - Christiana Care Health Services, Newark, Delaware
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan